CLINICAL TRIAL: NCT06864533
Title: Evaluation of Chemotherapy With Adjuvant Docetaxel After Radiotherapy for Localized High Malignant Prostate Cancer: A Prospective Muti-center Non-Randomized Controlled Trial
Brief Title: Adjuvant Chemotherapy for High Malignant Prostate Cancer
Acronym: PKUFH-GS5
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Collaborators: Peking University Shenzhen Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PKUFH-GS5
Record Dates: First submitted 2025-03-03; First posted 2025-03-07 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Prostate Cancer; Radiation Therapy; Chemotherapy; Gleason Score
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Docetaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Treatment Plus Chemotherapy Group (Experimental): This group will receive the standard radical treatment as in Arm 2, followed by adjuvant chemotherapy with docetaxel. Chemotherapy will start 4-8 weeks after the completion of radiotherapy. The chemotherapy regimen will consist of docetaxel 75 mg/m² administered intravenously on Day 1, repeated every 21 days for a total of 4-6 cycles. In cases of significant neuroendocrine differentiation and if well-tolerated, a combination of docetaxel and carboplatin (docetaxel 75 mg/m² and carboplatin AUC 4-6) will be used. Pre-treatment with dexamethasone will be administered to reduce potential side effects.
  Interventions: Drug: Docetaxel
- Standard Treatment Group (No Intervention): This group will receive the standard radical treatment for high-grade localized prostate cancer. Patients will undergo definitive or post operative radiotherapy. Endocrine therapy will be provided for high-risk patients as per NCCN guidelines, with a duration of 2 to 3 years with definitive radiotherapy . For postoperative patients, endocrine therapy will be given for salvage setting.

INTERVENTIONS:
Drug: Docetaxel — Chemotherapy will start 4-8 weeks after the completion of radiotherapy. The chemotherapy regimen will consist of docetaxel 75 mg/m² administered intravenously on Day 1, repeated every 21 days for a total of 4-6 cycles. In cases of significant neuroendocrine differentiation and if well-tolerated, a combination of docetaxel and carboplatin (docetaxel 75 mg/m² and carboplatin AUC 4-6) will be used. Pre-treatment with dexamethasone will be administered to reduce potential side effects.
  Other Names: carboplatin
  Arms: Standard Treatment Plus Chemotherapy Group

SUMMARY:
This study aims to evaluate the efficacy of adjuvant docetaxel chemotherapy following radical radiotherapy in patients with localized high-grade prostate cancer. Eligible participants include those diagnosed with prostate cancer confirmed by biopsy or surgical pathology, with a Gleason score of 9-10 or containing a Gleason 5 component, and no evidence of distant metastasis. Patients will be divided into two groups: the standard treatment group receiving only radical treatment (radiotherapy or surgery), and the standard treatment plus chemotherapy group, receiving four to six cycles of docetaxel chemotherapy after standard treatment. The primary endpoint is Failure-Free Survival (FFS), with secondary endpoints including Biochemical Relapse-Free Survival (BRFS), Metastasis-Free Survival (MFS), Overall Survival (OS), and assessment of adverse events The study aims to better understand the impact of adjuvant chemotherapy on the prognosis of patients with high-risk prostate cancer and determine whether it improves survival outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed prostate cancer diagnosed by biopsy or surgery with a Gleason score of 9-10 (GG grade 5) or containing Gleason 5 components.
2. No evidence of distant metastasis confirmed by imaging.
3. Expected to receive standard radical treatment or postoperative radiotherapy.
4. Estimated survival time greater than 12 months.
5. Aged ≥ 18 years.
6. Karnofsky Performance Status (KPS) ≥ 80.
7. Adequate blood count: white blood cell ≥ 3.5 × 10^9/L, neutrophils ≥ 1.5 × 10^9/L, platelets ≥ 100.0 × 10^

Exclusion Criteria:

1. History of malignant tumors (except those cured for more than 5 years).
2. Previous abdominal radiation therapy.
3. Weight loss > 10% within the past 6 months.
4. Pre-existing or concomitant bleeding disorders.
5. Active infections.
6. Significant cardiovascular disease (e.g., controlled hypertension, unstable angina, NYHA class ≥ II congestive heart failure, unstable symptomatic arrhythmias, or ≥ II peripheral vascular disease) or any condition deemed intolerable to chemotherapy by the oncology department.

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 315 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2031-09-01 (Estimated)

PRIMARY OUTCOMES:
Failure-Free Survivall，FFS | 5 years
  The time from radiotherapy to the first occurrence of any of the following events: biochemical relapse (defined as PSA rise meeting the criteria for biochemical recurrence), distant metastasis, or death.

SECONDARY OUTCOMES:
Biochemical relapse-free survival，BRFS | 5 years
  The time from radiotherapy to the first occurrence of biochemical relapse (defined as PSA rise meeting the criteria for biochemical recurrence)
Metastasis-free survival, MFS | 5 years
  The time from radiotherapy to the first occurrence of distant metastasis.
Overall survival, OS | 5 years
  The time from radiotherapy to the first occurrence of death.
Toxicities | 5 years
  The assessment of adverse events will be conducted using the Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Peking University Shenzhen Hospital, Shenzhen, Guangdong

IPD SHARING:
Plan to Share IPD: No